CLINICAL TRIAL: NCT01380119
Title: Phase 2 Study of Orally Formulated Heat-killed Mycobacterium Vaccae Study in TB Patients
Brief Title: Tuberculosis (TB) Immunotherapy Phase 2 Study
Acronym: imm02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lisichansk Regional Tuberculosis Dispensary (Other)
Collaborators: National Medical University, Ukraine (Other); Immunitor USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: imm02; LisichnskRTD (Other: LisichanskRTD)
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Tuberculosis
Keywords: sputum conversion; liver biochemistry; weight loss; quality of life
MeSH Terms: conditions — Tuberculosis; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- V7 (Experimental): Oral pill containing heat-killed Mycobacterium vaccae
  Interventions: Biological: V7
- Placebo pill (Placebo Comparator): Identically appearing placebo pills
  Interventions: Other: placebo

INTERVENTIONS:
Biological: V7 — experimental arm
  Arms: V7
Other: placebo — placebo pill
  Arms: Placebo pill

SUMMARY:
This is a phase II, randomized, placebo-controlled trial, aimed to seek the therapeutic benefit of V7 in combination with standard of care anti-Tuberculosis (TB) therapy (ATT) among Mycobacterium tuberculosis-infected sputum smear positive subjects. The results will be compared to placebo combined with standard ATT therapy. The trial will consist of one stage with sputum evaluation at months 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are at least 18 years old and are willing and capable of providing informed consent. Both men and non-pregnant women will be included.
* TB infection documented prior to Study Entry by sputum smear positive for acid-fast bacilli (AFB) test.
* TB score status at baseline.
* Agreement to participate in the study and to give a sample of blood for lab testing.
* Readily available home or other address where patient can be found.

Exclusion Criteria:

* Subjects who might have already taken V5 in prior trial and have no baseline data. Pregnant or breast-feeding women are excluded.
* Subjects who have taken study unrelated drugs or immunomodulatory therapies during study or prior to Entry.
* Medical conditions such as active alcohol or substance abuse, or psychological issues that in the opinion of the local investigator would interfere with adherence to the requirements of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
sputum conversion | 2 months
  To compare the efficacy of combination of V7 with anti-TB treatment versus anti-TB treatment+placebo in adults with pulmonary tuberculosis including:

SECONDARY OUTCOMES:
safety | 1 and 2 months
  1. Liver functions tests (AST and ALT, and bilirubin) as main biochemical tests
  2. To confirm quality of life improvement by specially designed questionnaire TB score
  3. The beneficial effect on TB-associated wasting by measuring body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Aldar Bourinbaiar, MD/PhD, Study Director — Immunitor USA Inc.
Locations (1):
- Lisichansk TB Dispensary, Lisichansk, Luhansk Oblast, Ukraine

REFERENCES:
- [Background] Arjanova OV, Prihoda ND, Yurchenko LV, Sokolenko NI, Frolov VM, Tarakanovskaya MG, Batdelger D, Jirathitikal V, Bourinbaiar AS. Adjunct oral immunotherapy in patients with re-treated, multidrug-resistant or HIV-coinfected TB. Immunotherapy. 2011 Feb;3(2):181-91. doi: 10.2217/imt.10.96. Epub 2010 Dec 24. PMID 21182457
- [Background] Arjanova OV, Prihoda ND, Yurchenko LV, Sokolenko NI, Vihrova LA, Pylypchuk VS, Frolov VM, Kutsyna GA. Enhancement of efficacy of tuberculosis drugs with Immunoxel (Dzherelo) in HIV-infected patients with active pulmonary tuberculosis. Immunotherapy. 2009 Jul;1(4):549-56. doi: 10.2217/imt.09.25. PMID 20635986
- [Background] Butov DA, Pashkov YN, Stepanenko AL, Choporova AI, Butova TS, Batdelger D, Jirathitikal V, Bourinbaiar AS, Zaitzeva SI. Phase IIb randomized trial of adjunct immunotherapy in patients with first-diagnosed tuberculosis, relapsed and multi-drug-resistant (MDR) TB. J Immune Based Ther Vaccines. 2011 Jan 18;9:3. doi: 10.1186/1476-8518-9-3. PMID 21244690
- [Result] Efremenko YV, Butov DA, Prihoda ND, Zaitzeva SI, Yurchenko LV, Sokolenko NI, Butova TS, Stepanenko AL, Kutsyna GA, Jirathitikal V, Bourinbaiar AS. Randomized, placebo-controlled phase II trial of heat-killed Mycobacterium vaccae (Longcom batch) formulated as an oral pill (V7). Hum Vaccin Immunother. 2013 Sep;9(9):1852-6. doi: 10.4161/hv.25280. Epub 2013 Jun 19. PMID 23782489
- [Result] Butov DA, Efremenko YV, Prihoda ND, Zaitzeva SI, Yurchenko LV, Sokolenko NI, Butova TS, Stepanenko AL, Kutsyna GA, Jirathitikal V, Bourinbaiar AS. Randomized, placebo-controlled Phase II trial of heat-killed Mycobacterium vaccae (Immodulon batch) formulated as an oral pill (V7). Immunotherapy. 2013 Oct;5(10):1047-54. doi: 10.2217/imt.13.110. PMID 24088075